CLINICAL TRIAL: NCT03274583
Title: Mobile Phone Detection of Atrial Fibrillation
Acronym: MODE-AF
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, University of Turku
Other Study IDs: T02/005/17
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: atrial fibrillation; smartphone; detection
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Patients being treated in the wards of Heart Center and Acute Internal Medicine of Turku University Hospital, Turku Finland between April and September 2017 with atrial fibrillation as the prevalent rhythm.
  Interventions: Diagnostic Test: Smartphone seismographic recording
- Control group: Patients being treated in the wards of Heart Center and Acute Internal Medicine of Turku University Hospital, Turku Finland between April and September 2017 with sinus rhythm as the prevalent rhythm.

INTERVENTIONS:
Diagnostic Test: Smartphone seismographic recording — A short recording of heart rhythm using a smartphone.
  Groups: Study Group

SUMMARY:
The aim of this study is to evaluate the reliability of smartphone seismocardiographic detection of AF in comparison to the gold standard of continuous telemetry ECG recording.

DETAILED DESCRIPTION:
In the this case-control study, 300 patients being treated in the wards of Heart Center and Department of Acute Internal Medicine of Turku University Hospital in Turku, Finland between April and September 2017 were included in the study. Patients were assigned to two groups according to the prevalent heart rhythm (sinus rhythm or atrial fibrillation). A smartphone equipped with an inbuilt accelerometer and a gyroscope was placed on the patient's chest to obtain a seismocardiographic recording. Simultaneous telemetry electrocardiography was obtained to assess the reliability of seismographic rhythm recordings. Results will be analyzed to describe the specificity and sensitivity of the method.

ELIGIBILITY:
Inclusion Criteria for patients with FA:

* ≥18 years of age
* telemetry ECG available
* being treated in Turku University Hospital Heart Center / Acute internal medicine ward
* atrial fibrillation

Inclusion Criteria for patients with sinus rhythm:

* ≥18 years of age
* telemetry ECG available
* being treated in Turku University Hospital Heart Center / Acute internal medicine ward
* sinus rhythm
* gender and age matching pair in FA group

Exclusion Criteria:

* ≤18 years of age
* paced rhythm
* cardioversion during preceding 7 days
* informed consent not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the wards of Heart Center and Acute Internal Medicine of Turku University Hospital, Turku Finland between April and September 2017.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of seismocardiography in diagnosing atrial fibrillation | 2017-2018

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Länsi-Suomen Lääni, Finland

IPD SHARING:
Plan to Share IPD: Undecided